CLINICAL TRIAL: NCT02701465
Title: Blood Flow - an Underlying Mechanism Behind Clinical Improvements in Patients With Subacromial Pain Syndrome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 666
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain
Keywords: Shoulder; Exercise therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The subjects in this arm will receive four high intensity (80% of peak work rate) four-minute interval exercises for the abduction movement in the plane of the scapula (m. supraspinatus), supervised three times per week. In addition they will perform the exercise program described for the control group.
  Interventions: Other: Exercise: local high intensity interval exercise
- Control group (Active Comparator): The control group will receive a best clinical practice home-exercise program, with regular follow-ups at the shoulder clinic every other week. The details are described in Granviken et al. (2015).
  Interventions: Other: Exercise: best clinical practice

INTERVENTIONS:
Other: Exercise: local high intensity interval exercise — The subjects in this arm will receive four high intensity (80% of peak work rate) four-minute interval exercises for the abduction movement in the plane of the scapula (m. supraspinatus), supervised three times per week. In addition they will perform the exercise program described for the control group.
  Arms: Intervention group
Other: Exercise: best clinical practice — The control group will receive a best clinical practice home-exercise program, with regular follow-ups at the shoulder clinic every other week. The details are described in Granviken et al. (2015).
  Arms: Control group

SUMMARY:
The purpose of this randomized clinical trial is two-fold. Firstly to see if patients suffering Subacromial Pain Syndrome can improve blood flow in the supraspinatus muscle in their shoulder, and secondly to investigate how changes in this blood flow are related to pain experience and shoulder function.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain for longer than three months
* clinical findings indicative of subacromial pain syndrome (evaluated by Hawkins-Kennedy sign, Neers sign, painful arch and Yokum test)
* normal passive range of motion of the shoulder

Exclusion Criteria:

* subjects unable to provide an informed consent
* lack of ability to complete the intervention
* full rupture of the tendon of m. supraspinatus
* planned shoulder surgery, or previous shoulder surgery on affected shoulder
* other musculoskeletal problem that could explain the symptoms
* adhesive capsulitis
* pregnancy
* rheumatoid arthritis
* symptomatic osteoarthritis of the shoulder/shoulder girdle
* glenohumeral instability
* widespread pain syndrome
* unstable underlying heart disease
* cortisone injections in the shoulder the last month
* allergies
* other serious mental or somatic disease (i.e. psychosis or active cancer disease).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Time to exhaustion, incremental test | Week 0
  participants abduct their shoulder up to 90 degrees in scapula's plane (scapularization) at a frequency of 0,5 Hz. Every minute the load is increased with 250 grams. The test is stopped if participant fails to maintain pace or movement quality, or experiences increased pain. Time at failure is noted as the result.

SECONDARY OUTCOMES:
SPADI questionnaire | Week 0
  Subjective pain and function outcomes (Likert scales)
SPADI questionnaire | Pre+post-test (8 weeks in-between)
  Subjective pain and function outcomes (Likert scales)
Weight | Week 0
  Weight (kg)
Height | Week 0
  Height (cm)
Age | Week 0
  Age (years)
Duration of symptoms | Week 0
  Duration of symptoms (months)
Affected shoulder | Week 0
  What shoulder is affected (left/right)
Socioeconomic status | Week 0
  The patient fills in a questionnaire stating number of children, marital status, welfare status and working situation
1 repetition maximum (1RM), bilateral shoulder test | Week 0
  After warmup: maximal strength was measured as the weight the subject could manage to lift once - usually achieved in 3-5 attempts. The movement conducted was the earlier described scapularization movement.
1 repetition maximum (1RM), bilateral shoulder test | Week 8
  After warmup: maximal strength was measured as the weight the subject could manage to lift once - usually achieved in 3-5 attempts. The movement conducted was the earlier described scapularization movement.
Time to exhaustion, steady state | Week 0
  Subject abduct their shoulder up to 90 degrees in scapula's plane (scapularization) at a frequency of 0,5 Hz. The load is set to 80% of the incremental time to exhaustion test. The test is stopped if the fails to maintain pace or movement quality, or the subject experience increased pain. Time at failure is noted as the result.
Time to exhaustion, steady state | Week 8
  Subject abduct their shoulder up to 90 degrees in scapula's plane (scapularization) at a frequency of 0,5 Hz. The load is set to 80% of the incremental time to exhaustion test. The test is stopped if the fails to maintain pace or movement quality, or the subject experience increased pain. Time at failure is noted as the result.
Regional blood flow in m. supraspinatus, using contrast enhanced ultrasound (concentration of white analyzed as decibels in region of interest) | Week 0
  Baseline images will be taken with ultrasonic device to confirm an intact m. supraspinatus. An intravenous line will be inserted in the contralateral arm and the patient will be injected with a bolus of contrast dye (Optison, 3 ml bolus, 0.19 mg / mL perflutren). The injection is administered by a physician related to the research project. Measurements of regional blood flow at rest made are of the supraspinatus tendon. Then the participants perform a standardized training exercise to recruit the vasculature in m. supraspinatus (scapularization to 90 degrees, 80% of TTU weight (incremental), 3 minutes). Post-exercise images are taken immediately after this.
Regional blood flow in m. supraspinatus, using contrast enhanced ultrasound (concentration of white analyzed as decibels in region of interest) | Week 8
  Baseline images will be taken with ultrasonic device to confirm an intact m. supraspinatus. An intravenous line will be inserted in the contralateral arm and the patient will be injected with a bolus of contrast dye (Optison, 3 ml bolus, 0.19 mg / mL perflutren). The injection is administered by a physician related to the research project. Measurements of regional blood flow at rest made are of the supraspinatus tendon. Then the participants perform a standardized training exercise to recruit the vasculature in m. supraspinatus (scapularization to 90 degrees, 80% of TTU weight (incremental), 3 minutes). Post-exercise images are taken immediately after this.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hoff, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, back-neck-shoulder multidiciplinary clinic, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No